CLINICAL TRIAL: NCT02391545
Title: A Two-arm, Phase 1b/2 Study of Duvelisib Administered in Combination With Rituximab or Obinutuzumab in Subjects With Previously Untreated CD20+ Follicular Lymphoma (CONTEMPO)
Brief Title: A Study of Duvelisib in Combination With Rituximab or Obinutuzumab in Subjects With Previously Untreated CD20+ Follicular Lymphoma (CONTEMPO)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor is focusing on studies which can enable registration of duvelisib.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-19; 2014-005459-13 (EudraCT Number)
Record Dates: First submitted 2015-03-03; First posted 2015-03-18 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: CD20+ Follicular Lymphoma
Keywords: Follicular Lymphoma; Previously Untreated
MeSH Terms: conditions — Lymphoma, Follicular | interventions — duvelisib; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duvelisib and Rituximab (Experimental): Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  Interventions: Drug: Duvelisib; Drug: Rituximab
- Duvelisib and Obinutuzumab (Experimental): Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Obinutuzumab 1000 mg will be administered intravenously (IV) beginning at Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  Interventions: Drug: Duvelisib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Duvelisib — PI3K Inhibitor
  Other Names: Copiktra, IPI-145
Drug: Rituximab — monoclonal antibody
  Other Names: Rituxan/MabThera®
  Arms: Duvelisib and Rituximab
Drug: Obinutuzumab — monoclonal antibody
  Other Names: GAZYVA/GAZYVARO™
  Arms: Duvelisib and Obinutuzumab

SUMMARY:
A Two-arm, Phase 1b/2 Study of duvelisib Administered in Combination with Rituximab or Obinutuzumab in Subjects with Previously Untreated CD20+ Follicular Lymphoma.

DETAILED DESCRIPTION:
This is a two-arm, open-label, Phase 1b/2 trial designed to evaluate the safety and efficacy of duvelisib in combination with rituximab and duvelisib in combination with obinutuzumab in subjects with previously untreated CD20+ FL.

The study will be conducted in two parts, a Safety Lead-in (Part 1) followed by a randomized, 2-Stage Design in Part 2. Each treatment arm will be assessed independently for dose limiting toxicity (DLT) within Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20+, follicular lymphoma that has not been treated
* CD20-immunophenotyping of tumor to document B-cell follicular lymphoma
* Stage II disease with bulky disease (≥ 7cm lesion), Stage III, or Stage IV disease
* Disease that requires treatment based on the Investigator's opinion (e.g., meets GELF criteria)
* At least one measurable lesion that is > 1.5 cm in at least one dimension
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (corresponds to Karnofsky Performance Status [KPS] >=60%)

Exclusion Criteria:

* Received systemic treatment for lymphoma such as chemotherapy, immunotherapy, radiotherapy, investigational agents, or radioimmunotherapy.
* Clinical evidence of transformation to a more aggressive subtype of lymphoma or grade 3B follicular lymphoma
* Severe allergic or anaphylactic reaction to any monoclonal antibody therapy, murine protein, or known hypersensitivity to any of the study drugs
* Prior allogeneic hematopoietic stem cell transplant
* Prior, current or chronic hepatitis B or hepatitis C infection
* Human immunodeficiency virus (HIV) infection or Human T Cell Lymphotropic Virus 1 (HTLV-1) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-17 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (21):
- United States (5):
  - Los Angeles, California
  - Palo Alto, California
  - Hackensack, New Jersey
  - Rochester, New York
  - Dallas, Texas
- Belgium (3):
  - Kortrijk
  - Leuven
  - Wilrijk
- France (5):
  - Clermont-Ferrand
  - Marseille
  - Pessac
  - Rouen
  - Tours
- Italy (2):
  - Bologna
  - Varese
- Spain (4):
  - Badalona, Barcelona
  - Barcelona
  - Madrid
  - Salamanca
- United Kingdom (2):
  - Leeds
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Duvelisib and Obinutuzumab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Obinutuzumab 1000 mg will be administered intravenously (IV) beginning at Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  IPI-145 (duvelisib): PI3K Inhibitor
  Obinutuzumab
- Duvelisib and Rituximab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  IPI-145 (duvelisib): PI3K Inhibitor
  Rituximab
Period: Overall Study
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Started | 27 | 28
Completed | 1 | 0
Not Completed | 26 | 28
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Termination of study by sponsor | 20 | 20
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other Reasons | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 20 | 36
  >=65 years | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.32) | 58.2 (10.65) | 58.3 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 11 | 18 | 29
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 3 | 9
  United States | 10 | 9 | 19
  United Kingdom | 3 | 2 | 5
  Italy | 1 | 1 | 2
  France | 3 | 4 | 7
  Spain | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLTs) - Part 1
Time Frame: 28 days from first dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Duvelisib and Obinutuzumab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Obinutuzumab 1000 mg will be administered intravenously (IV) beginning at Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  Duvelisib: PI3K Inhibitor
  Obinutuzumab
- Duvelisib and Rituximab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. IPI-145 will be administered orally, twice daily, in 28-day cycles.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  Duvelisib: PI3K Inhibitor
  Rituximab
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 27 | 28
Participants | 1 | 0

2. Primary Outcome: Complete Response Rate (CRR)- Part 2
Time Frame: Up to 2 years from the first dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 27 | 28
Participants | 11 | 10

3. Secondary Outcome: Safety: Composite Measure of Safety, as Indicated by Treatment-emergent Adverse Events (TEAEs) and Changes in Safety Laboratory Values
Description: Composite measure of safety, as indicated by Treatment-emergent adverse events (TEAEs) and changes in safety laboratory values. TEAEs assessed as >=Grade 3.
Time Frame: Up to 30 days after the last dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Duvelisib and Rituximab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules. Duvelisib will be administered orally, twice daily, in 28-day cycles.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Cycle 1 (28 day cycles); days 1, 8, 15 and 22. Thereafter, infusions will occur on Day 1 of the even cycles treatment; Cycles 4-26.
  Duvelisib: PI3K Inhibitor
  Rituximab
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 27 | 28
Participants
  TEAEs assessed as ≥ Grade 3 | 24 | 19
  TEAEs ≥ Grade 3 assessed as related to duvelisib | 23 | 17
  TEAEs ≥ Grade 3 assessed as related to anti-CD20 | 11 | 2

4. Secondary Outcome: Overall Response Rate (ORR)
Time Frame: Up to 2 years from the first dose of study treatment
Measure: Number; unit: participants
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 27 | 28
participants
  Complete Response | 11 | 10
  Partial Response | 13 | 16
  Stable Disease | 1 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: The median DOR was non-estimable.
Time Frame: Up to 2 years from the first dose of study treatment
Population: Data could not be reported because the study was terminated early and a sufficient number of subjects and events were not available for analysis.
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 2 years from the first dose of study treatment
Population: The study had been terminated and Overall Survival was not performed.
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetic (PK): Plasma Concentrations of Duvelisib and IPI-656 (Metabolite)
Description: Plasma concentrations of Duvelisib and IPI-656 (metabolite)
Time Frame: Every 4 weeks for 16 weeks
Population: The study had been terminated and PK analysis was not performed.
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 35 months
Arm/Group | Duvelisib and Obinutuzumab | Duvelisib and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/28
Serious Adverse Events (participants affected / at risk) | 16/27 | 10/28
Other Adverse Events (participants affected / at risk) | 26/27 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib and Obinutuzumab (N=27) | Duvelisib and Rituximab (N=28)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 2
Fatigue (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Conjuctivitis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia respiratory synctial viral (Infections and infestations) | 1 | 0
Pylonephritis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia Cytomegaloviral (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib and Obinutuzumab (N=27) | Duvelisib and Rituximab (N=28)
Neutropenia (Blood and lymphatic system disorders) | 5 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 12 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 16
Abdominal Pain (Gastrointestinal disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 4 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 8 | 9
Pyrexia (General disorders) | 8 | 6
Asthenia (General disorders) | 4 | 5
Malaise (General disorders) | 4 | 1
Mucosal Inflammation (General disorders) | 2 | 3
Chills (General disorders) | 1 | 2
Drug Hypersensitivity (Immune system disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1
Conjuctivitis (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 13 | 9
Aspartate aminotransferase increased (Investigations) | 13 | 8
Amylase increased (Investigations) | 3 | 3
Lipase increased (Investigations) | 3 | 3
Transaminases increased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 4 | 4
Dizziness (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 3 | 5
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Orthostatic Hypotension (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes